CLINICAL TRIAL: NCT05738447
Title: A Phase I Study of mRNA Vaccine for Patients With HBV-positive Advanced Hepatocellular Carcinoma
Brief Title: Application of mRNA Immunotherapy Technology in Hepatitis B Virus-related Refractory Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Xingchen Peng, Professor, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-1371
Record Dates: First submitted 2023-01-30; First posted 2023-02-22 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Liver Cancer; Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; mRNA vaccine; HBV; immunotherapy
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Cohort (Experimental): With 20ug as the starting point, the dose was increased using a dose escalation scheme. Each subject only received one corresponding dose, and the intramuscular injection was administered again every 7 days, and after 4 doses, the 5th dose was given after 1-month interval.
  Interventions: Biological: HBV mRNA vaccine

INTERVENTIONS:
Biological: HBV mRNA vaccine — With 20ug as the starting point, the dose was increased using a dose escalation scheme. Each subject only received one corresponding dose, and the intramuscular injection was administered again every 7 days, and after 4 doses, the 5th dose was given after 1-month interval.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of mRNA vaccine for HBV-positive Advanced Hepatocellular Carcinoma.

DETAILED DESCRIPTION:
Hepatocellular carcinoma is a common malignant tumor of the digestive system worldwide and is particularly prevalent in China. More than 80% of hepatocellular carcinoma patients in China have concomitant hepatitis B virus infection. However, there are limited effective treatments for hepatocellular carcinoma that have failed standard treatment, and the prognosis for these patients is poor. About 350 million people worldwide are chronically infected with the hepatitis B virus (HBV), and chronic HBV infection accounts for at least 50% of hepatocellular carcinoma cases worldwide. Therefore, anti-HBV can be a potential target for hepatocellular carcinoma.

The mRNA vaccines are a highly promising novel anti-tumor approach. The applicant team of this project has carried out research on raw materials and preparation process, vaccine stability, quality standard, delivery vector construction, and anti-tumor mechanism of action of mRNA immune formulation in the early stage. Now we have completed the optimized design of mRNA raw materials, and the construction and optimization of the mRNA delivery vector. The tumor therapeutic mRNA immune formulation with high efficiency, safety, scalable preparation, and quality control has been selected and preclinical evaluation has been completed to verify its safety and efficacy. The project has constructed mRNA vaccines, and no similar therapeutic method or product has been reported in the international arena.

This project proposes to conduct a phase I clinical study based on the previous study to include patients with advanced hepatocellular carcinoma who have failed second-line standard treatment or cannot receive standard treatment. A dose-escalation trial will be conducted, and one effective dose will be selected for a fixed-dose trial to explore the safety, tolerability, and efficacy of mRNA immunotherapy technology for clinical application. Project implementation is expected to benefit a wide range of hepatocellular carcinoma patients and improve their prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients: ≥ 18 years old; ≤ 70 years old;
2. Patients with HBV-positive advanced hepatocellular carcinoma after failure of second-line standard therapy (including PD-1 inhibitor therapy, chemotherapy, and anti-vascular targeted drugs);
3. HBsAg positive, regardless of whether the peripheral blood is positive for HBV DNA.
4. ECOG physical fitness score: 0~1 points;
5. Estimated survival ≥ 3 months;
6. The main organs have good function, that is, the relevant examination indicators within random 14 days meet the following requirements:

   1. Blood routine examination: hemoglobin ≥ 80 g/L (no blood transfusion within 14 days); Neutrophil count> 1.5×109/L; Platelet count≥ 80×109/L;
   2. Biochemical examination: total bilirubin ≤ 1.5× ULN (upper limit of normal); alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤ 2.5×ULN; If liver metastases are present, ALT or AST ≤ 5×ULN; Endogenous creatinine clearance

      ≥ 60 ml/min (Cockcroft-Gault formula);
   3. Cardiac Doppler ultrasound assessment: left ventricular ejection fraction (LVEF) ≥50%.
7. Sign the informed consent form;
8. Good compliance, family members agree to cooperate with survival follow-up.

Exclusion Criteria:

1. Participated in clinical trials of other drugs within 4 weeks;
2. The patient has a history of other tumors, unless it is cervical cancer in situ, treated cutaneous squamous cell carcinoma or bladder epithelial tumor or other malignant tumors that has received radical treatment (at least 5 years before enrollment)
3. Patients with uncontrolled cardiac clinical symptoms or diseases, such as heart failure above NYHA grade 2, unstable angina, myocardial infarction within 1 year, and clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention.
4. For female subjects: pregnant or lactating women.
5. The patient has active tuberculosis, bacterial or fungal infection (≥ grade 2 of NCI-CTC, 3rd edition); There is HIV infection with active HBV infection, HCV infection.
6. Those who have a history of psychotropic drug abuse and have mental disorders that cannot be remitted;
7. The subject has any active autoimmune disease or has a history of autoimmune disease (such as, but not limited to uveitis, enteritis, pituitary inflammation, nephritis, hyperthyroidism, hypothyroidism; Participants with vitiligo or who had complete remission of asthma in childhood and did not require any intervention in adulthood could be included; Participants in asthma requiring medical intervention with bronchodilators omitted).
8. According to the judgment of the investigator, there are concomitant diseases that seriously endanger the safety of patients or affect the completion of the patient's research.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2023-02-15 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Adverse events | up to 12 months
  Adverse events defined as the number of participants with adverse events according
Objective response rate | up to 12 months
  ORR is defined as the percentage of patients who achieve a response, which can either be complete response (complete disappearance of lesions) or partial response (reduction in the sum of maximal tumor diameters by at least 30% or more)
Progress-Free Survival | up to 12 months
  PFS is defined as the time from the administration of the first dose to first disease
Overall Survival | up to 12 months]
  OS is defined as the time from the administration of the first dose to death

CONTACTS AND LOCATIONS:
Overall Officials: Xingchen Peng, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Zhang BH, Yang BH, Tang ZY. Randomized controlled trial of screening for hepatocellular carcinoma. J Cancer Res Clin Oncol. 2004 Jul;130(7):417-22. doi: 10.1007/s00432-004-0552-0. PMID 15042359
- [Background] Ganem D, Prince AM. Hepatitis B virus infection--natural history and clinical consequences. N Engl J Med. 2004 Mar 11;350(11):1118-29. doi: 10.1056/NEJMra031087. No abstract available. PMID 15014185
- [Background] Parkin DM. The global health burden of infection-associated cancers in the year 2002. Int J Cancer. 2006 Jun 15;118(12):3030-44. doi: 10.1002/ijc.21731. PMID 16404738
- [Background] Mittal S, El-Serag HB. Epidemiology of hepatocellular carcinoma: consider the population. J Clin Gastroenterol. 2013 Jul;47 Suppl(0):S2-6. doi: 10.1097/MCG.0b013e3182872f29. PMID 23632345
- [Background] Chang MH, Chen CJ, Lai MS, Hsu HM, Wu TC, Kong MS, Liang DC, Shau WY, Chen DS. Universal hepatitis B vaccination in Taiwan and the incidence of hepatocellular carcinoma in children. Taiwan Childhood Hepatoma Study Group. N Engl J Med. 1997 Jun 26;336(26):1855-9. doi: 10.1056/NEJM199706263362602. PMID 9197213
- [Background] Greenberg DP. Pediatric experience with recombinant hepatitis B vaccines and relevant safety and immunogenicity studies. Pediatr Infect Dis J. 1993 May;12(5):438-45. doi: 10.1097/00006454-199305000-00037. PMID 8327313
- [Background] Liaw YF, Sung JJ, Chow WC, Farrell G, Lee CZ, Yuen H, Tanwandee T, Tao QM, Shue K, Keene ON, Dixon JS, Gray DF, Sabbat J; Cirrhosis Asian Lamivudine Multicentre Study Group. Lamivudine for patients with chronic hepatitis B and advanced liver disease. N Engl J Med. 2004 Oct 7;351(15):1521-31. doi: 10.1056/NEJMoa033364. PMID 15470215
- [Background] Papatheodoridis GV, Lampertico P, Manolakopoulos S, Lok A. Incidence of hepatocellular carcinoma in chronic hepatitis B patients receiving nucleos(t)ide therapy: a systematic review. J Hepatol. 2010 Aug;53(2):348-56. doi: 10.1016/j.jhep.2010.02.035. Epub 2010 Apr 27. PMID 20483498
- [Background] Papatheodoridis GV, Chan HL, Hansen BE, Janssen HL, Lampertico P. Risk of hepatocellular carcinoma in chronic hepatitis B: assessment and modification with current antiviral therapy. J Hepatol. 2015 Apr;62(4):956-67. doi: 10.1016/j.jhep.2015.01.002. Epub 2015 Jan 13. PMID 25595883
- [Background] Isogawa M, Chung J, Murata Y, Kakimi K, Chisari FV. CD40 activation rescues antiviral CD8(+) T cells from PD-1-mediated exhaustion. PLoS Pathog. 2013;9(7):e1003490. doi: 10.1371/journal.ppat.1003490. Epub 2013 Jul 11. PMID 23853599
- [Background] Virgin HW, Wherry EJ, Ahmed R. Redefining chronic viral infection. Cell. 2009 Jul 10;138(1):30-50. doi: 10.1016/j.cell.2009.06.036. PMID 19596234
- [Background] Shouval D, Roggendorf H, Roggendorf M. Enhanced immune response to hepatitis B vaccination through immunization with a Pre-S1/Pre-S2/S vaccine. Med Microbiol Immunol. 2015 Feb;204(1):57-68. doi: 10.1007/s00430-014-0374-x. Epub 2015 Jan 4. PMID 25557605
- [Background] Nishikawa J, Yoshiyama H, Iizasa H, Kanehiro Y, Nakamura M, Nishimura J, Saito M, Okamoto T, Sakai K, Suehiro Y, Yamasaki T, Oga A, Yanai H, Sakaida I. Epstein-barr virus in gastric carcinoma. Cancers (Basel). 2014 Nov 7;6(4):2259-74. doi: 10.3390/cancers6042259. PMID 25386788
- [Background] Reinhard K, Rengstl B, Oehm P, Michel K, Billmeier A, Hayduk N, Klein O, Kuna K, Ouchan Y, Woll S, Christ E, Weber D, Suchan M, Bukur T, Birtel M, Jahndel V, Mroz K, Hobohm K, Kranz L, Diken M, Kuhlcke K, Tureci O, Sahin U. An RNA vaccine drives expansion and efficacy of claudin-CAR-T cells against solid tumors. Science. 2020 Jan 24;367(6476):446-453. doi: 10.1126/science.aay5967. Epub 2020 Jan 2. PMID 31896660
- [Background] Wang F, Qin Z, Lu H, He S, Luo J, Jin C, Song X. Clinical translation of gene medicine. J Gene Med. 2019 Jul;21(7):e3108. doi: 10.1002/jgm.3108. Epub 2019 Jul 15. PMID 31246328
- [Background] Fenton OS, Kauffman KJ, McClellan RL, Kaczmarek JC, Zeng MD, Andresen JL, Rhym LH, Heartlein MW, DeRosa F, Anderson DG. Customizable Lipid Nanoparticle Materials for the Delivery of siRNAs and mRNAs. Angew Chem Int Ed Engl. 2018 Oct 8;57(41):13582-13586. doi: 10.1002/anie.201809056. Epub 2018 Sep 14. PMID 30112821
- [Background] Miao L, Li L, Huang Y, Delcassian D, Chahal J, Han J, Shi Y, Sadtler K, Gao W, Lin J, Doloff JC, Langer R, Anderson DG. Delivery of mRNA vaccines with heterocyclic lipids increases anti-tumor efficacy by STING-mediated immune cell activation. Nat Biotechnol. 2019 Oct;37(10):1174-1185. doi: 10.1038/s41587-019-0247-3. Epub 2019 Sep 30. PMID 31570898
- [Background] Hou X, Zhang X, Zhao W, Zeng C, Deng B, McComb DW, Du S, Zhang C, Li W, Dong Y. Author Correction: Vitamin lipid nanoparticles enable adoptive macrophage transfer for the treatment of multidrug-resistant bacterial sepsis. Nat Nanotechnol. 2020 Jul;15(7):615. doi: 10.1038/s41565-020-0675-8. PMID 32346117